CLINICAL TRIAL: NCT01215799
Title: A Phase II Study of Bafetinib (INNO-406) as Treatment for Patients With Hormone-Refractory Prostate Cancer
Brief Title: Study of Bafetinib (INNO-406) as Treatment for Patients With Hormone-Refractory Prostate Cancer
Acronym: PROACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAFETINIB-P2-HRPC-01
Record Dates: First submitted 2010-09-30; First posted 2010-10-07 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Hormone Refractory Prostate Cancer; HRPC
MeSH Terms: interventions — bafetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bafetinib (Experimental)
  Interventions: Drug: Bafetinib

INTERVENTIONS:
Drug: Bafetinib — Bafetinib 240 mg bid
  Other Names: INNO-406

SUMMARY:
This is a Phase II open-label study evaluating the preliminary efficacy and safety of bafetinib administered as 240 mg orally twice daily in subjects with Hormone Refractory Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males age ≥18 years.
* Histologically confirmed diagnosis of adenocarcinoma of the prostate.
* Hormone-refractory prostate cancer having progressed despite androgen deprivation therapy that resulted in a castrated level of testosterone (<50 ng/dL) or orchiectomy; with or without evidence of measurable or evaluable disease.
* PSA increase defined as 2 consecutive rises; first increase in PSA occurred a minimum of 1 week from the reference value; increase in PSA should be at least 25% above the reference value and absolute PSA value should be >5 ng/mL.
* May have received no more than 1 prior chemotherapy regimen. Prior immunomodulatory therapy (sipuleucel-t (Provenge), interferon) is allowed.
* Must be taking a single agent LHRH agonist or antagonist, unless previously underwent orchiectomy.
* ECOG performance status 0-2.
* Able to swallow pills.
* Able to provide written, voluntary informed consent, comply with trial procedures, and have accessibility to the site.

Exclusion Criteria:

* Chemotherapy, antibody therapy, major surgery or irradiation within 4 weeks of study enrollment
* Exposure to any investigational agent within 30 days of the Screening Visit.
* No prior flutamide (Eulexin) and ketoconazole use within 4 weeks, bicalutamide (Casodex) within 6 weeks or nilutamide (Nilandron) within 6 weeks of study enrollment.
* Use of Quadramet therapy during 2 months prior to study enrollment or Metastron ever.
* Prior treatment with a tyrosine kinase inhibitor.
* Subjects who have started bisphosphonate therapy within 4 weeks of study enrollment are excluded. Subjects treated with a stable dose of a bisphosphonate for >4 weeks and the tumor has still progressed can be enrolled in the study.
* Known CNS disease or CNS metastases.
* History of other malignancies within the last five years except curatively treated basal cell carcinoma or superficial bladder cancer.
* Laboratory values: Screening serum creatinine greater than or equal to 1.5 x ULN, alanine aminotransferase (ALT) greater than 3 times the upper limit of normal, total bilirubin greater than 3 times the upper limit of normal, white blood cell (WBC) count <3500/mm3, absolute neutrophil count <1500/mm3, hematocrit level <35% and platelets <100,000/mm3.
* History of abnormal bleeding or use of anticoagulant therapy.
* Clinically evident congestive heart failure >class II of the New York Heart Association (NYHA) guidelines.
* Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
* History of MI within 6 months or uncontrolled angina within 3 months.
* Severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, chronic renal disease, chronic liver disease.
* Known HIV infection.
* Uncontrolled active, infection.
* Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
* Any condition that in the opinion of the Investigator is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | At six months.
  The primary objective of this study is to determine the preliminary efficacy of administration of bafetinib in subjects with hormone-refractory prostate cancer (HRPC), as measured by the objective response rate (ORR), which is a combination of CR (PSA ≤0.12 ng/mL) and PR (≥50% reduction in PSA from baseline).

SECONDARY OUTCOMES:
Safety | At six months.
  The safety of bafetinib in this population assessed by the frequency and severity of adverse events (AEs), abnormal findings on physical examination, laboratory tests, and vital signs.
Progression-free survival | At six months.
  Progression-free survival is defined as the time from enrollment to first documentation of objective PSA or tumor progression, or to death due to any cause in the absence of previous documentation of objective tumor progression.
Objective tumor response | At six months.
  The total proportion of subjects who have an objective tumor reponse (CR + PR) using the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Levitt, M.D., Ph.D., Study Director — Chief Medical Officer, CytRx Corporation
Locations (1):
- City of Hope Medical Center, Duarte, California, United States